CLINICAL TRIAL: NCT06297603
Title: A Phase 3, Randomized, Multicenter, Double-Blind Study to Investigate the Efficacy and Safety of Retatrutide Once Weekly Compared With Placebo in Adult Participants With Type 2 Diabetes, Moderate or Severe Renal Impairment With Inadequate Glycemic Control on Basal Insulin With or Without Metformin and/or SGLT2 Inhibitor
Brief Title: Effect of Retatrutide Compared With Placebo in Participants With Type 2 Diabetes and Moderate or Severe Renal Impairment, With Inadequate Glycemic Control on Basal Insulin, With or Without Metformin and/or SGLT2 Inhibitor (TRANSCEND-T2D-3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18806; J1I-MC-GZQA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Kidney Disease; Renal Insufficiency Chronic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus; Kidney Diseases; Renal Insufficiency, Chronic | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide administered subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide administered SC.
  Interventions: Drug: Retatrutide
- Retatrutide Dose 3 (Experimental): Participants will receive retatrutide administered SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2; Retatrutide Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of retatrutide compared with placebo in participants with Type 2 Diabetes and renal impairment, with inadequate glycemic control on basal insulin alone or a combination of basal insulin with or without metformin and/or sodium-glucose cotransporter-2 (SGLT2) inhibitor. The study will last about 14 months and may include up to 22 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥7.0% (53 millimoles per mole (mmol/mol)) to ≤10.5% (91 mmol/mol)
* Have moderate or severe renal impairment
* Have been on the following stable diabetes treatment during 90 days prior to screening

  * basal insulin (≥20 International Units (IU)/day) with or without
  * metformin and/or SGLT2 inhibitor
* Are of stable weight for at least 90 days prior to screening
* Have a Body Mass Index (BMI) ≥23.0 kilograms per meter squared (kg/m2)

Exclusion Criteria:

* Have Type 1 Diabetes (T1D)
* Have a history of ketoacidosis or hyperosmolar state or coma within the last 6 months prior to screening
* Have a history of severe hypoglycemia or hypoglycemia unawareness within the last 6 months prior to screening
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have a history of unstable or rapidly progressing renal disease
* Have a prior or planned surgical treatment for obesity
* Have New York Heart Association Functional Classification III or IV congestive heart failure
* Have had acute myocardial infarction, stroke, or were hospitalized for congestive heart failure within 90 days prior to screening
* Have a known clinically significant gastric emptying abnormality
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) syndrome Type 2.
* Have any lifetime history of a suicide attempt
* Had chronic or acute pancreatitis
* Have taken prescribed or over-the-counter medication, or alternative remedies, intended to promote body weight reduction within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) (%) | Baseline, Week 52

SECONDARY OUTCOMES:
Percentage of Participants Achieving HbA1c <7.0% | Week 52
Percentage of Participants Achieving HbA1c ≤6.5% | Week 52
Change from Baseline in Fasting Serum Glucose | Baseline, Week 52
Percentage of Time Continuous Glucose Monitoring (CGM) Glucose Values are Between 70 and 180 mg/dL | Week 52
  Measured during the CGM session that occurs during 30 days prior to Week 52
Percent Change from Baseline in Body Weight | Baseline, Week 52
Change from Baseline in Body Weight | Baseline, Week 52
Percentage of Participants Achieving Weight Reduction of ≥5% | Week 52
Percentage of Participants Achieving Weight Reduction of ≥10% | Week 52
Percentage of Participants Achieving Weight Reduction of ≥15% | Week 52
Percentage of Participants Achieving HbA1c ≤6.5% and ≥10% Weight Reduction | Week 52
Percent Change from Baseline in Non-HDL Cholesterol | Baseline, Week 52
Percent Change from Baseline in Triglycerides | Baseline, Week 52
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (28):
  - Nephrology Consultants, Huntsville, Alabama
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Kidney & Hypertension Center - Apple Valley, Apple Valley, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - EndoTrials Center for Clinical Research, La Mesa, California
  - UCLA South Bay Endocrinology, Torrance, California
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Orita Clinical Research, Decatur, Georgia
  - CARE Institute, Idaho Falls, Idaho
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Billings Clinic, Billings, Montana
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - NYC Research INC, Long Island City, New York
  - Research Foundation of SUNY - University of Buffalo, Williamsville, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Central States Research, Tulsa, Oklahoma
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Prime Revival Research Institute, LLC, Flower Mound, Texas
  - Juno Research, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah
- Argentina (17):
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - CEDIC, CABA
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Centro Médico Colón, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - CIMeL, Lanús
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - DIM Clínica Privada, Ramos Mejía
  - INECO Neurociencias Oroño, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
- Brazil (7):
  - Centro de Diabetes Curitiba, Curitiba
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Praxis Pesquisa Medica, Santo André
  - Instituto de Pesquisa Clinica, São Paulo
  - CEDOES, Vitória
- Israel (7):
  - Clalit Health Services - Atlit, Atlit
  - Soroka Medical Center, Beersheba
  - Institute of Diabetes, Technology and Research - Clalit Health, Herzliya
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
- Mexico (4):
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Medical Care and Research SA de CV, Mérida
  - FAICIC S. de R.L. de C.V., Veracruz
- Puerto Rico (3):
  - Centro de Endocrinologia Alcantara Gonzalez, Bayamón
  - Isis Clinical Research Center, Guaynabo
  - Mgcendo Llc, San Juan
- United Kingdom (9):
  - Southmead Hospital, Bristol
  - Edinburgh Royal Infirmary, Edinburgh
  - Panthera Biopartners - Glasgow, Glasgow
  - George Eliot Hospital, Nuneaton
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Salford Royal Hospital, Salford
  - Lister Hospital, Stevenage
  - The Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Effect of Retatrutide Compared With Placebo in Participants With Type 2 Diabetes and Moderate or Severe Renal Impairment, With Inadequate Glycemic Control on Basal Insulin, With or Without Metformin and/or SGLT2 Inhibitor (TRANSCEND-T2D-3) — https://trials.lilly.com/en-US/trial/466881